CLINICAL TRIAL: NCT00370149
Title: A Randomized, Controlled Trial of Catheter Related Infectious Event Rates Using Antibiotic-impregnated Catheters vs. Conventional Catheters in Pediatric Cardiovascular Surgery Patients
Brief Title: Study of Catheter-related Infections Using Antibiotic-coated Versus Conventional Catheters in Children
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Blinded interim analysis resulted in early termination of the study.
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0512-37
Record Dates: First submitted 2006-08-28; First posted 2006-08-30 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-01

CONDITIONS: Infection Prevention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antibiotic-impregnated Catheters (M/R) (Active Comparator): Interventions is insertion intra-operatively of catheters impregnated with minocycline and rifampin to determine if their is a therapeutic difference between this catheter and the placebo (non-impregnated) catheter. The catheters are sized to accommodate children in different size ranges: Cook Inc. Double Lumen 4 Fr., 8 cm long, (C-UDLM-401J-ABRM-HC), 5 Fr., 8 cm long, (C-UDLM-501J-ABRM-HC), and 5 Fr., 12 cm long, (C-UDLMY-501J-RSC-ABRM-HC).
  Interventions: Device: Antibiotic-impregnated Catheters (M/R)
- Non-impregnated Catheter (C/S) (Placebo Comparator): Intervention is insertion intra-operatively of conventional, non-impregnated catheters. There are two sizes to accommodate children in different size ranges: Cook Incorporated Double Lumen Polyurethane Central Venous Catheters, 4 Fr., 8 cm long, (C-UDLM-401J), 5 Fr., 8 cm long, (C-UDLM-501J), and 5 Fr., 12 cm long (C-UDLM-501J-RSC).
  Interventions: Device: Non-impregnated Catheters (C/S)

INTERVENTIONS:
Device: Antibiotic-impregnated Catheters (M/R) — Patients randomized to this arm will have the antibiotic-impregnated catheters inserted intra-operatively. The catheters are sized to accommodate children in different size ranges.
  Arms: Antibiotic-impregnated Catheters (M/R)
Device: Non-impregnated Catheters (C/S) — Patients randomized to this arm will have the central venous catheter inserted intra-operatively. The catheters are sized to accommodate children in different size ranges.
  Arms: Non-impregnated Catheter (C/S)

SUMMARY:
The primary purpose of the study is to determine if a therapeutic difference exists between central venous catheters impregnated with minocycline and rifampin and conventional catheters not impregnated with antibiotics when used in children at high risk for bloodstream infections (CABSI) after cardiac surgery.

DETAILED DESCRIPTION:
The standard central venous catheter (CVC) is now commonly used for infants, children, and adults. The antibiotic-coated CVC is a newer CVC gaining popularity for use in adults. The Food and Drug Administration (FDA) and the Center for Disease Control (CDC) support use of the antibiotic-coated CVC for adult patients. But the FDA and CDC have not yet endorsed use of the antibiotic-coated CVC for infants and children due to lack of research on this CVC in infants and children.

ELIGIBILITY:
Inclusion Criteria:

* Age < 18 years
* Cardiovascular surgery patient with a case complexity warranting CVC placement longer than 3 days
* Study devices of appropriate size for patient use without modification
* Informed consent obtained prior to patient entering the operating room

Exclusion Criteria:

* Age ≥ 18 years
* Drug allergy to minocycline, other tetracyclines, or rifampin
* Ventricular assist device (VAD) therapy
* Extracorporeal membrane oxygenation (ECMO) therapy
* Patients undergoing cardiac transplant
* Any active infection or being treated for bacteremia at the time of randomization

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 326 (Actual)
Dates: Start 2006-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine G. Cox, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cox EG, Knoderer CA, Jennings A, Brown JW, Rodefeld MD, Walker SG, Turrentine MW. A Randomized, Controlled Trial of Catheter-Related Infectious Event Rates Using Antibiotic-Impregnated Catheters Versus Conventional Catheters in Pediatric Cardiovascular Surgery Patients. J Pediatric Infect Dis Soc. 2013 Mar;2(1):67-70. doi: 10.1093/jpids/pis066. Epub 2012 Jul 4. PMID 26619445

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and consented during pre-operative visits at Riley Hospital between September 2006 and May 2010. Study catheters were assigned a random identification number by Cook Critical Care, Bloomington, IN. The clinical and infection control teams were blinded to which arm a patient was assigned.
Pre-assignment Details: Patients <18 years of age who had cardiovascular surgery with a case complexity warranting a central venous catheter received either an antibiotic impregnated catheter or a conventional non-impregnated catheter on a randomized, blinded 1:1 ratio.
Groups:
- Antibiotic Impregnated Catheters (M/R): Randomization to the 2 arms of the study were on a blinded a 1:1 allocation. Patients randomized to M/R had the catheter impregnated with minocycline and rifampin (M/R) inserted intraoperatively. The specific Central Venous Catheters are the Cook Incorporated Spectrum Double Lumen Polyurethane Central Venous Catheters, 4 Fr., 8 cm long, (C-UDLM-401J-ABRM), 5 Fr., 8 cm long, (C-UDLM-501J-ABRM-HC), and 5 Fr., 12 cm long, (C-UDLMY-501J-RSC-ABRM).
- Conventional Non-impregnated Catheters (C/S): Randomization to 2 arms of the study were on a blinded a 1:1 allocation. Patients randomized to this arm had the conventional Central Venous Catheter (C/S) with no antibiotic coating inserted intraoperatively. The specific catheters are the Cook Incorporated Double Lumen Polyurethane Central Venous Catheters, 4 Fr., 8 cm long, (C-UDLM-401J), 5 Fr., 8 cm long, (C-UDLM-501J), and 5 Fr., 12 cm long, (C-UDLM-501J-RSC).
Period: Overall Study
Arm/Group | Antibiotic Impregnated Catheters (M/R) | Conventional Non-impregnated Catheters (C/S)
Started | 165 | 161
Completed | 146 | 142
Not Completed | 19 | 19
Not completed — Physician Decision | 16 | 16
Not completed — Protocol Violation | 1 | 0
Not completed — Catheter inserted in wrong vessel- | 2 | 1
Not completed — Pre-existing infection | 0 | 1
Not completed — Antibiotic coated dressing placed | 0 | 1

BASELINE CHARACTERISTICS:
Population: Patients <18 years of age who had cardiovascular surgery with a case complexity warranting a central venous catheter received either an antibiotic impregnated catheter or a conventional non-impregnated catheter on a randomized, blinded 1:1 ratio.
Groups:
- Antibiotic Impregnated Catheters (M/R): Patients randomized to this arm had the M/R inserted intra-operatively as determined by the blinded randomization procedure (1M/R: 1C/S). The catheters were sized to accommodate children in different size ranges: Cook Incorporated Spectrum Double Lumen Polyurethane Central Venous Catheters, 4 Fr., 8 cm long, (C-UDLM-401J-ABRM) and C-UDLM-401J-ABRM-HC), 5 Fr., 8 cm long, (C-UDLM-501J-ABRM-HC), and 5 Fr., 12 cm long, (C-UDLMY-501J-RSC-ABRM-HC).
- Conventional Non-impregnated Catheters (C/S): Patients randomized to this arm had the C/S inserted intra-operatively as determined by the blinded randomization procedure (1M/R: 1 C/S). The catheters were one of two sizes to accommodate children in different size ranges: Cook Incorporated Double Lumen Polyurethane Central Venous Catheters,4 Fr., 8 cm long, (C-UDLM-401J), 5 Fr., 8 cm long, (C-UDLM-501J), or 5 Fr., 12 cm long, (C-UDLM-501J RSC).
- Total: Total of all reporting groups
Arm/Group | Antibiotic Impregnated Catheters (M/R) | Conventional Non-impregnated Catheters (C/S) | Total
Number analyzed (Participants) | 165 | 161 | 326
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 165 | 161 | 326
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 84 | 168
  Male | 81 | 77 | 158
Region of Enrollment [Number; unit: participants]
  United States | 165 | 161 | 326

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Catheter-related Bloodstream Infections (CRBSI) Per 1000 Catheter Days
Description: Rates of CRBSI defined as 1. micro-organism isolated from a blood culture; 2. Clinical manifestations of infection such as fever (≥38 C) and/or hypotension (defined according to age-related practice guidelines for systolic blood pressure); 3. No apparent source for the bloodstream infection except for the catheter.
Time Frame: Participants were followed for the duration of the hospital stay, an average of 6 days.
Population: The intention-to-treat population consisted of all randomized participants with valid informed consent. Participants were analyzed according to the treatment assigned at randomization.
Measure: Number; unit: participants
Groups:
- Antibiotic Impregnated Catheters (M/R): Patients randomized to this arm had the M/R inserted intra-operatively as determined by the blinded randomization procedure (1M/R: 1C/S). The catheters were one of two to accommodate children in different size ranges: Cook Incorporated Spectrum Double Lumen Polyurethane Central Venous Catheters, 4 Fr., 8 cm long, (C-UDLM-401J-ABRM), 5 Fr. 8 cm long, (C-UDLM-501J-ABRM-HC), or 5 Fr., 12 cm long, (C-UDLMY-501J-RSC-ABRM).
- Conventional Non-impregnated Catheters (C/S): Patients randomized to this arm had the C/S inserted intra-operatively as determined by the blinded randomization procedure (1M/R: 1 C/S). The catheters were one of two to accommodate children in different size ranges: Cook Incorporated Double Lumen Polyurethane Central Venous Catheters,4 Fr., 8 cm long, (C-UDLM-401J), 5 Fr., 8 cm long, (C-UDLM-501J), or 5 Fr., 12 cm long, (C-UDLM-501J-RSC).
Arm/Group | Antibiotic Impregnated Catheters (M/R) | Conventional Non-impregnated Catheters (C/S)
Number analyzed (Participants) | 146 | 142
participants | 3 | 3

2. Secondary Outcome: Episodes of Clinical Sepsis and/or Infection With Identified Source Other Than Catheter
Description: A secondary outcome measure was episodes of clinical sepsis and/or infection with identified source other than the CVC.
Time Frame: Participants were followed for the duration of hospital stay, an average of 6 days.
Population: The intention-to-treat population consisted of all randomized participants with valid informed consent. Participants were analyzed according to treatment assigned at randomization.
Measure: Number; unit: participants
Groups:
- Antibiotic Impregnated Catheters (M/R): Patients randomized to this arm had the M/R inserted intra-operatively as determined by the blinded randomization procedure (1M/R: 1C/S). The catheters were one of two sizes to accommodate children in different size ranges: Cook Incorporated Spectrum Double Lumen Polyurethane Central Venous Catheters, 4 Fr., 8 cm long, (C-UDLM-401J-ABRM), ), 5 Fr., 8 cm long, (C-UDLM-501J-ABRM-HC) or 5 Fr., 12 cm long, (C-UDLMY-501J-RSC-ABRM).
- Conventional Non-impregnated Catheters (C/S): Patients randomized to this arm had the C/S inserted intra-operatively as determined by the blinded randomization procedure (1M/R: 1 C/S). The catheters were one of two sizes to accommodate children in different size ranges: Cook Incorporated Double Lumen Polyurethane Central Venous Catheters,4 Fr., 8 cm long, (C-UDLM-401J), 5 Fr., 8 cm long, (C-UDLM-501J), 5 Fr., 12 cm long, (C-UDLM-501J-RSC).
Arm/Group | Antibiotic Impregnated Catheters (M/R) | Conventional Non-impregnated Catheters (C/S)
Number analyzed (Participants) | 146 | 142
participants | 8 | 4

3. Secondary Outcome: Death
Description: Patient Death during hospitalization.
Time Frame: Participants were followed for the duration of the hospital stay, an average of 6 days.
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- Conventional Non-impegnated Catheters (C/S): Patients randomized to this arm had the C/S inserted intra-operatively as determined by the blinded randomization procedure (1M/R: 1 C/S). The catheters were one of two sizes to accommodate children in different size ranges: Cook Incorporated Double Lumen Polyurethane Central Venous Catheters,4 Fr., 8 cm long, (C-UDLM-401J), 5 Fr., 8 cm long, (C-UDLM-501J) 5 Fr.,12 cm long, (C-UDLM-501J-RSC).
Arm/Group | Antibiotic Impregnated Catheters (M/R) | Conventional Non-impegnated Catheters (C/S)
Number analyzed (Participants) | 146 | 142
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse device effects and adverse events were collected during the participants' hospitalizations which ranged from 5 - 10 days.
Description: Daily evaluation through hospital discharge included fever, blood pressure, white blood cell count, platelet count, glucose, arrhythmia, urine output, or additional antibiotic administration. Any catheter related complication, including pneumothorax, thrombosis,occlusion, displacement, leakage, fracture, or fragmentation was recorded.
Groups:
- Antibiotic Impregnated Catheters (M/R): Randomization to the 2 arms of the study were on a blinded a 1:1 allocation with the objective of determining if a therapeutic difference existed between M/R and C/S catheters. Patients randomized to this Arm had the M/R catheter inserted intra-operatively. Patients receiving this Catheter were enrolled in the study. The specific CVCs are the Cook Incorporated Spectrum Double Lumen Polyurethane Central Venous Catheters, 4 Fr., 8 cm long, (C-UDLM-401J-ABRM), 5 Fr., 8 cm long, (C-UDLM-501J-ABRM-HC), and 5 Fr., 12 cm long, (C-UDLMY-501J-RSC-ABRM-HC). Patients were followed for adverse device affects and adverse events through their hospitalization stay.
- Conventional Non-impregnated Catheters (C/S): Randomization to 2 arms of the study were on a blinded a 1:1 allocation with the objective of determining if there was a therapeutic difference between the M/R and C/S catheters. Patients randomized to this arm had the C/S inserted intra-operatively. Patients receiving this catheter were enrolled in the study.The specific catheters are the Cook Incorporated Double Lumen Polyurethane Central Venous Catheters, 4 Fr., 8 cm long, (C-UDLM-401J), 5 Fr., 8 cm long, (C-UDLM-501J), 5 Fr., 12 cm long, (C-UDLM-501J-RSC). Patients were followed for adverse device affects and adverse events through their hospitalization stay
Arm/Group | Antibiotic Impregnated Catheters (M/R) | Conventional Non-impregnated Catheters (C/S)
Serious Adverse Events (participants affected / at risk) | 1/146 | 1/142
Other Adverse Events (participants affected / at risk) | 7/146 | 10/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antibiotic Impregnated Catheters (M/R) (N=146) | Conventional Non-impregnated Catheters (C/S) (N=142)
Electromechanical Disassociation resulting in death (Cardiac disorders) | 1 (1) | 0 (0)
Respiratory Failure and Chronic lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antibiotic Impregnated Catheters (M/R) (N=146) | Conventional Non-impregnated Catheters (C/S) (N=142)
Other Catheter related Complications (Infections and infestations) | 7 (7) | 10 (10)

LIMITATIONS AND CAVEATS:
A blinded interim analysis by an independent Data Safety Monitoring Board resulted in early termination of the study: of 288 evaluable patients, the rates of CRBSI and line-related complications were similar between the 2 groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No